CLINICAL TRIAL: NCT04970355
Title: Efficacy of Erenumab in Chronic Cluster Headache: A 10 Week Double-blind, Randomized, Placebo Controlled, Multicentric Trial.
Brief Title: Efficacy of Erenumab in Chronic Cluster Headache
Acronym: CHERUB01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Uwe Reuter, Neurologist, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CAMG334ADE07T; 2020-004399-16 (EudraCT Number)
Record Dates: First submitted 2021-07-11; First posted 2021-07-21 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Cluster Headache; Trigeminal Autonomic Cephalalgias; Headache Disorders, Primary; Brain Disease
Keywords: Pain; Neurology
MeSH Terms: conditions — Cluster Headache; Trigeminal Autonomic Cephalalgias; Headache Disorders, Primary; Brain Diseases; Pain | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Erenumab (Experimental): Double-Blind Treatment Phase: Participants receive erenumab 280 mg subcutaneous (SC) injections (loading dose, week 0) followed by erenumab 140 mg s.c. in week 4.
  Interventions: Biological: Erenumab
- Placebo (Placebo Comparator): Double-Blind Treatment Phase: Participants receive placebo subcutaneous (SC) injections in week 0 and week 4.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Erenumab — Pre-filled syringe; s.c. injection
  Other Names: AMG 334
  Arms: Erenumab
Drug: Placebo — Pre-filled syring; s.c. injection
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy of erenumab in participants with chronic cluster headache.

DETAILED DESCRIPTION:
The purpose of this study is to determine the efficacy of erenumab in a loading dose of 280mg followed by 140mg after 4 weeks compared to placebo as a prophylactic treatment in patients with chronic cluster headache.

This study has a 10-week 2-arm, randomized, double-blind, parallel- group, placebo-controlled design. Data from this study will provide important information if the blockade of the CGRP receptor with erenumab is an efficacious principle for the treatment of chronic cluster headache

ELIGIBILITY:
Inclusion Criteria (screening)

* Adults ≥18 and < 65 years of age
* Documented history of chronic cluster headache for ≥12 months prior to screening according to the International Classification of Headache Disorders-3rd Edition (ICHD-3)
* Participants are able to distinguish cluster headache attacks from other headaches.
* Insufficient efficacy OR tolerability OR contraindications of approved cluster headache prophylactic medications. Insufficient efficacy and tolerability as determined by the patient.
* Sufficient acute attack treatment with triptans or oxygen based on the patient´s history
* The patient is able to distinguish cluster headache attacks from other headaches (i.e. tension-type headaches).

Inclusion Criteria (Baseline)

* At least 9 cluster headache attacks as defined by the ICHD-3 in 7 days during the baseline epoch (SPII), confirmed by patient-reported eDiary entries.
* Attacks must have occurred on more than 50% of days of the baseline epoch (SPII).
* ≥ 90% patient-reported eDiary compliance during the Baseline epoch, compliance is measured as interacting with e-Diary at least once a day.

Exclusion Criteria:

* Diagnosis or history of other primary headache diseases according to the International Classification of Headache Disorders, 3rd Edition (ICHD-3), excluding episodic tension type headache and migraine as defined in criterion 2.
* Headache freedom from the historic diagnosis of migraine has to be at least one year prior to study inclusion. If patients have on average <=1 migraine attack per month within a year and can distinguish between migraine attacks and cluster attacks, they are allowed to participate.
* Unable to differentiate cluster headache attacks from other headaches
* Use of a prophylactic cluster headache medication within 5 half-lives prior to the start of the baseline phase
* Parallel use of an SPG stimulator, deep brain stimulation or parallel use of a device for the acute/preventive treatment of chronic cluster headache
* Administration of botulinum toxin type A or B in the head or neck area, within 4 months of baseline (SP II)
* Concurrent use of other therapeutic monoclonal antibodies.
* Current use or any prior exposure to any calcitonin-gene-related peptide (CGRP) antibody, any antibody to the CGRP receptor
* Use of other investigational drugs within 5 half-lives of enrollment, or until the expected pharmacodynamic effect has returned to baseline, whichever is longer
* Evidence of drug, opioid or alcohol abuse or dependence within 12 months prior to screening, based on medical records or patient self-report
* History of use of psilocybin (mushrooms), LSD, MDMA or 2- bromo-LSD within 2 months prior to baseline (SPII)
* Have a positive urine drug screen (UDS) for any substances of abuse, except cannabis or cannabinoids, prior to randomization. A retest is applicable if, in judgment of the investigator, there is a reasonable explanation for the positive result. A negative result in the retest is obligatory for entering baseline (SPII)
* Diagnosis or history of significant active or unstable psychiatric disease, such as bipolar disorder, schizophrenia, personality disorders, or other serious mood or anxiety disorders. Patients with anxiety disorder and/or major depressive disorder are permitted in the study if they are considered by the investigator to be stable and are taking no more than one medication per disorder. Patients must have been on a stable dose within the 3 months prior to the start of the baseline phase
* Score "yes" on item 4 or item 5 of the Suicidal Ideation section of the Columbia Suicide Severity Rating Scale (C-SSRS), if this ideation occurred in the past month, or "yes" on any item of the Suicidal Behavior section, except for the "Non-Suicidal Self-Injurious Behavior" (item also included in the Suicidal Behavior section), if this behavior occurred in the past 3 months. Patients who do not meet this criterion, but who are considered by the judgment of the investigator to be at significant risk for suicide, must be excluded
* Active chronic pain syndromes (e.g., fibromyalgia or chronic pelvic pain) in which the pain has lost its guiding and warning function and has acquired an independent disease value.
* History or current evidence of major psychiatric disorder (such as schizophrenia, bipolar disorder or type B personality disorder that might interfere with the ability to properly report clinical outcomes)
* History or current severe coronary artery disease, myocardial infarction, stroke, transient ischemic attack, unstable angina, or coronary artery bypass surgery or other revascularization procedures within 12 months prior to screening
* History or current diagnosis of ECG abnormalities indicating significant risk of safety for patients participating in the study- Known hypersensitivity to multiple drugs, monoclonal antibodies or other therapeutic protein
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases
* Hepatic disease by history or total bilirubin ≥2×ULN or ALT or AST ≥3xULN as assessed by central laboratory at initial screening
* History of severe constipation, defined as less than 3 bowel movements /week not adequately manageable by routine medical treatment, within 3 months prior to screening
* Acute SARS-CoV2 Infection within 2 weeks prior to screening
* Women who are pregnant or nursing
* Known hypersensitivity to multiple drugs, monoclonal antibodies or other therapeutic proteins, or to erenumab or to any of the inactive ingredients
* Unlikely to be able to complete all protocol required study visits or procedures, and/or to comply with all required study procedures (e.g., independent completion of electronic diary items) to the best of the patient's and investigator's knowledge
* Prior known treatment with a CGRP receptor mAb (erenumab)
* Prior treatment with a CGRP ligand antibody. Exceptions: Patients who participated in a randomized, placebo-controlled trial with CGRP ligand antibodies and were not unblinded (i.e., have no knowledge whether they received placebo or verum) can participate in the trial. Patients, who knowingly received a CGRP ligand antibody (i.e.galcanezumab or fremanezumab) can participate in the trial if the following criteria are met: a) Administered dose was not effective versus placebo in clinical trials i.e. galcanezumab (<300 mg/month s.c.) or fremanezumab (≤675 mg loading dose followed by 225 mg s.c./month), b) Treatment duration of maximal 2 month or 2 injection cycles c) The last dose was administered at least 6 month prior to begin of screening epoche.
* Patients who may be dependent on the sponsor or investigator
* Patients who are in custody of an institution due to governmental authority decision or court order

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Reduction of weekly cluster headache attack frequency from baseline over the last 2 weeks of the double-blind epoch (averaged for 7 days). | Baseline; Weeks 5-6 (Days 29-42)
  Number of cluster headache attacks was recorded daily by study participants in their ePRO Diary, Baseline and 6 weeks of daily data during double-blind treatment phase will be converted into 7-calendar day intervals: The baseline 7-10 day interval, Week 5+6.

SECONDARY OUTCOMES:
Percentage of participants with a 50% or greater reduction from baseline in the weekly number of cluster headache attacks averaged per 7 days over the last 2 weeks of the DB epoch. | Baseline; Weeks 5-6 (Days 29-42)
  A 50% responder is any participant who has a ≥50% reduction from baseline in the weekly number of cluster headache attacks in a 7-day interval: Weeks 5+6
Patient Global Impression of Improvement (PGI-I) at week 6. | Baseline; Week 6
  PGI-I requests participants to mark the box that best describes their cluster headache condition since they started taking the medicine. The options in the displayed boxes are represented on a 7-point scale, with 1 = very much better, 2 = much better, 3 = a little better, 4 = no change, 5 = a little worse, 6 = much worse, and 7 = very much worse.

OTHER OUTCOMES:
Reduction from baseline in the weekly number of CH attacks in each of the last 2 weeks of the double blind epoch. | Baseline, Week 5; Week 6
  Number of cluster headache attacks was recorded daily by study participants in their ePRO Diary, Baseline and 6 weeks of daily data during double-blind treatment phase will be converted into 7-calendar day intervals: The baseline 7-10 day interval, week 5 and week 6.
Reduction from baseline in the number of weekly CH attacks over the entire double-blind trial period (day 1-42). | Baseline, Weeks 1- 6
  Number of cluster headache attacks was recorded daily by study participants in their ePRO Diary, Baseline and 6 weeks of daily data during double-blind treatment phase will be converted into 7-calendar day intervals: The baseline 7-10 day interval; week 1-week 6
Safety and tolerability of erenumab/placebo | Baseline; Week 1-Week 10
  Number of AEs, TEAEs, SAEs, and number of patients discontinue study participation stratified for treatment and non-treatment related discontinuation.
Discontinuation of the study due to intolerable attack frequency or severity during the double-blind epoch of the study. | Baseline; Week 1-Week 6
  To compare erenumab with placebo in reduction of frequency and intensity of CH attacks assessed by the rate of patients discontinuing the study due to intolerable attack frequency or severity.
Number of patients achieving at least a 30% reduction from baseline in weekly CH attacks averaged over the last 2 weeks (days 29-42) of the double-blind epoch | Baseline, Week 5-Week 6
  A 30% responder is any participant who has a ≥30% reduction from baseline in the weekly number of cluster headache attacks in a 7-day interva in Weeks 5+6
Number of patients achieving at least a 70 % reduction from baseline in weekly CH attacks averaged over the last 2 weeks (days 29-42) of the double-blind epoch. | Baseline, Week 5-Week 6
  A 70% responder is any participant who has a ≥70% reduction from baseline in the weekly number of cluster headache attacks in a 7-day interval: Weeks 5+6
Change from baseline in SF-12 quality of life at week 6 (day 42). Difference between erenumab and placebo scores at week 6 | Baseline; Week 6
  This information will help keep track of how participants feel and how well they are able to do usual activities.
Change from baseline in HIT-6 quality of life at week 6 (day 42). Difference between erenumab and placebo scores at week 6 and improvement of HIT-6 scores from baseline. | Baseline; Week 6
  This information will allow to assess the impact of attacks on headache related disability. The recall period for 3 questions is 4weeks & the remaining questions do not have a specific recall period.
Change from baseline in average duration in minutes of recorded CH attacks over the last 2 weeks (days 29-42) of the double-blind epoch. | Baseline: Weeks 5-6
  Duration of CH attacks was recorded daily by study participants in their ePRO Diary, Baseline and 6 weeks of daily data during double-blind treatment phase will be converted into 7-calendar day intervals: The baseline 7-10 day interval, Week 5+6.
Change from baseline in frequency of acute medication per week averaged over week 5 and 6 (days 29-42). | Baseline: Weeks 5-6
  Baseline data and the mean change from baseline in the overall weekly average number of days with the use of cluster-specific acute headache medications (as liosted in the protocoll) during weeks 5-6 after administration of the first dose of study drug (based on Week 0 to 5-6 data) is reported.
Change from baseline in average intensity in average numerical pain rating scale value of recorded attacks over week 5 and 6 (days 29-42). | Baseline: Weeks 5-6
  Participants marked the level of CH-associated pain using the numerical pain ratiung scale.
Discontinuation of treatment due to all-cause during the double-blind epoch of the study | Weeks 1-8
  Rate of patients discontinuing treatment due to any cause during the double-blind treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Reuter, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (11):
- Germany (11):
  - LMU Klinikum München, München, Bavaria
  - Kopfschmerzzentrum Frankfurt, Frankfurt am Main, Hesse
  - Vitos - Orthopädische Klinik gGmbH, Kassel, Hesse
  - Universitätsmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Universitätsklinikum Rostock, Rostock, Mecklenburg-Vorpommern
  - Praxis für Neurologie, Nervenheilkunde, Psychosomatik, Essen, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinik Dresden, Dresden, Saxony
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
  - Schmerzklinik Kiel - Migräne- und Kopfschmerzzentrum, Kiel, Schleswig-Holstein
  - Charité Universitätsmedizin Berlin, Berlin

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: CSR
Time Frame: Data are available 6 months after the primary publication.
Access Criteria: A research proposal must be approved by Charité Universitätsmedizin Berlin. Researchers must sign a data sharing agreement.

REFERENCES:
- [Derived] Mecklenburg J, Gaul C, Fitzek M, Overeem LH, Heinze A, Fleischmann R, Boeger A, Holle-Lee D, Straube A, Gendolla A, Israel-Willner H, Lorenz M, Gossrau G, Naegel S, Rimmele F, Rattan S, Materne B, Schulze D, Raffaelli B, Reuter U; CHERUB01 Study Group. Erenumab for Chronic Cluster Headache: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jun 2;8(6):e2516318. doi: 10.1001/jamanetworkopen.2025.16318. PMID 40526384